CLINICAL TRIAL: NCT04375124
Title: Evaluation of the Possible Role of Angiotensin Peptide (1-7) on Treatment of COVID-19
Brief Title: Treatment of Angiotensin Peptide (1-7) for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hasan Onal, Professor, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSSEAH--0059
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Biological Products

STUDY DESIGN:
Intervention Model Description: This group will receive angiotensin peptide (1-7) during their treatment at hospital.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-peptide group (No Intervention): This group will receive routine treatment and care for COVID-19.
- peptide group (Active Comparator): This group will receive angiotensin peptide (1-7) supplementation in addition to routine treatment and care for COVID-19.
  Interventions: Biological: Biological/Vaccine: Angiotensin peptide (1-7) derived plasma

INTERVENTIONS:
Biological: Biological/Vaccine: Angiotensin peptide (1-7) derived plasma — angiotensin peptide (1-7) derived plasma will be given to COVID-19 positive participants
  Arms: peptide group

SUMMARY:
Novel Coronavirus is reported to cause COVID-19, recently. It's known that this virus uses ACE (angiotensin converting enzyme) 2 receptors to enter human cells and also blocks the activity of ACE 2. Upon these data the investigators hypothesize that, mortal hyper-inflammation state which is shown in COVID-19 cases, can be a result of angiotensin peptide (1-7) deficiency. Therefore, the aim of this study is to evaluate the possible effect of angiotensin peptide (1-7) supplementation on treatment of COVID-19 cases.

DETAILED DESCRIPTION:
Novel Coronavirus is reported to cause COVID-19, recently. It's known that this virus uses ACE (angiotensin converting enzyme) 2 receptors to enter human cells and also blocks the activity of ACE 2. Upon these data the investigators hypothesize that, mortal hyper-inflammation state which is shown in COVID-19 cases, can be a result of angiotensin peptide (1-7) deficiency. Therefore, the aim of this study is to evaluate the possible effect of plasma derived angiotensin peptide (1-7) supplementation on treatment of COVID-19 cases.

ELIGIBILITY:
Inclusion Criteria:

* accepted to participate with an informed consent
* proven positive COVID-19

Exclusion Criteria:

* declined to participate
* genetic/chromosomal abnormalities
* any kind of history of previous adverse events with transfusion
* diagnosis of immune deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
mortality | 4 months
  mortality rates in two groups will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided